CLINICAL TRIAL: NCT00003428
Title: Phase II Randomized Double-Blind Evaluation of Two Dose Levels of LY353381 Hydrochloride Administered to Women With Locally Advanced or Metastatic Breast Cancer
Brief Title: Hormone Therapy in Treating Women With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 98-038; CDR0000066453 (Registry Identifier: PDQ (Physician Data Query)); LILLY-H4Z-MC-JWWD(a); NCI-G98-1451
Record Dates: First submitted 1999-11-01; First posted 2004-09-13 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Drug: arzoxifene hydrochloride

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using arzoxifene hydrochloride may fight breast cancer by blocking the use of estrogen by the tumor cells.

PURPOSE: This randomized phase II trial is comparing two different doses of arzoxifene hydrochloride to see how well it works in treating women with advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the response rate or clinical benefit rate in patients with locally advanced or metastatic breast cancer treated with 1 of 2 different doses of arzoxifene hydrochloride. II. Compare the response rates and clinical benefit rates for patients with tamoxifen-sensitive versus tamoxifen-refractory disease. III. Compare the degree of toxicity between the 2 doses of arzoxifene hydrochloride in these patients. IV. Compare the quality of life and survival of these patients receiving high versus low dose arzoxifene hydrochloride. V. Determine the time to progressive disease, time to treatment failure, and response duration of this treatment in these patients. VII. Measure changes in serum estradiol, follicle stimulating hormone, luteinizing hormone, and sex hormone binding globulin in these patients during treatment.

OUTLINE: This is a randomized, double blind study. Patients are stratified according to number of metastatic sites (less than 3 vs 3 or more), tamoxifen sensitivity (sensitive vs refractory), and degree of estrogen receptor positivity (high vs low vs unknown). Patients are randomized to receive 1 of 2 doses of arzoxifene hydrochloride. Patients receive arzoxifene hydrochloride orally once daily for 12 weeks. Treatment continues in the absence of toxicity and disease progression. Quality of life is assessed before, during, and at the completion of the study. Patients are followed every 4 weeks for 12 weeks, at 30 days after the last treatment, and every 2-3 months after the last treatment.

PROJECTED ACCRUAL: This study will accrue 104-114 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven locally advanced or metastatic breast cancer and meeting one of the following criteria: No prior systemic therapy OR Relapsed more than 12 months after stopping adjuvant tamoxifen (tamoxifen- sensitive) OR Relapsed while receiving adjuvant tamoxifen for more than 12 months (tamoxifen-refractory) OR Disease progression while receiving tamoxifen as first-line treatment for metastatic breast cancer (tamoxifen-refractory) Evaluable or bidimensionally measurable disease No rapid disease progression requiring chemotherapy Brain metastases allowed if stable for at least 6 months after surgery or radiotherapy, with no increase in corticosteroids Hormone receptor status: Estrogen receptor positive AND/OR Progesterone receptor positive OR Unknown status allowed if over 50 years old

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Female Menopausal status: Not specified Performance status: ECOG 0-1 Life expectancy: At least 24 weeks Hematopoietic: Granulocyte count at least 1500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL, transfusion independent Hepatic: Bilirubin no greater than 1.5 times normal PT/PTT no greater than 1.25 times upper limit of normal (ULN) ALT/AST no greater than 2.5 times ULN Renal: Creatinine less than 1.5 times ULN Calcium no greater than 11 mg/dL No hypercalcemia Other: Not pregnant or nursing Fertile patients must use approved nonhormonal contraceptive during and for 3 months after study No known predisposition to thromboembolic disorder At least 5 years since other primary malignancy except: Adequately treated nonmelanomatous skin cancer Carcinoma in situ of the cervix No serious concurrent systemic disorders incompatible with study

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Concurrent hematopoietic growth factor allowed Chemotherapy: No prior chemotherapy for metastatic breast cancer No concurrent chemotherapy Endocrine therapy: No prior hormonal therapy for metastatic breast cancer (except tamoxifen) No concurrent supplemental estrogen or progesterone At least 3 weeks since prior estrogen replacement therapy No other concurrent hormone therapy Radiotherapy: At least 2 weeks since prior radiotherapy Surgery: Not specified Other: At least 4 weeks since prior use of other investigational agents Concurrent bisphosphonate therapy allowed No other concurrent investigational agent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 1998-05; Primary Completion 2001-06 (Actual); Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifford A. Hudis, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States